CLINICAL TRIAL: NCT06544317
Title: Motor Intervention for Children With Developmental Coordination Disorder
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zhiguang Ji (Other)
Responsible Party: Sponsor-Investigator, Zhiguang Ji, doctor, Shanghai University of Medicine and Health Sciences
Organization: Shanghai University of Medicine and Health Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ShanghaiUMHS
Record Dates: First submitted 2024-07-19; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Developmental Coordination Disorder
MeSH Terms: conditions — Motor Skills Disorders | interventions — Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- training group (Experimental)
  Interventions: Behavioral: physical training
- control group (No Intervention)
- typically developing (Active Comparator)
  Interventions: Behavioral: physical training

INTERVENTIONS:
Behavioral: physical training — All children received a series of 90-minute sessions 3 times a week for 8 weeks of after-school physical training. Each session began with a warm-up (20 min), three or four tasks related to the skill to be developed (aerobic training, resistance training, other activities designed to improve motor skills and balance, stretching and flexibility activities and core strength and posture exercises; 60 min) and a cool-down (10 min). Children were divided into six groups, with the number of children in each group ranging from eight to twelve.
  Arms: training group; typically developing

SUMMARY:
This study focuses on the effects of physical activity in schools on the cognitive function and physical fitness of children with and without developmental coordination disorder (DCD). Methods: 58 children with DCD participated in an 8-week exercise program. Children's standing broad jump (SBJ), 50m dash, 50m*8 shuttle run, mental rotation and executive functions were assessed before and after training. A mixed-design analysis of variance (ANOVA) was conducted separately for each performance variable.

DETAILED DESCRIPTION:
Potential children were identified from elementary schools in three districts of Shanghai. The study protocol was approved by the Ethics Committee of Shanghai Uni-versity of Medicine and Health Sciences. In order to select the research sample, recruitment letters were sent to the parents of all children; these letters detailed the purpose, significance and research process of the study, and a consent form was attached. If parents were willing to participate in the study, they were asked to sign the consent form and scan the QR code to fill in the questionnaire, including DCDQ, the Attention Deficit/Hyperactivity Disorder (ADHD) Rating Scale-VI and other personal information. All questionnaire contents were only accessible to research team members, and the researcher's name and telephone number were provided in case parents had questions. A total of 2,761 children and their parents volunteered to participate in this study. Children were screed using the Developmental Coordination Disorder Questionnaire (DCDQ) . Teachers selected those children with probable DCD but without any intellectual or cognitive impairment. These children were then tested using the Movement Assessment Battery for Children, 2nd edition. Finally, 116 pDCD children were randomly divided into a training group (TG, mean age 10.67 ± 1.25 years, 50 boys and 8 girls) and a control group (CG, mean age 10.27 ± 1.04 years, 48 boys and 10 girls) and gender matched typically developing (TD, mean age 10.35 ± 1.87 years; 48 boys and 12 girls) controls were included in the study. TG and TD will receive an additional 8 weeks of physical training intervention, while CG will not participate in the physical training intervention.

ELIGIBILITY:
Inclusion Criteria:

* DCDQ scores as follows: (8-9 years: < 56 points; 10-12 years: < 58 points)
* one subitem of the MABC-2 rank below 15%
* age 9 to 11 years old (elementary school age)

Exclusion Criteria:

* Children with other mental illness who are unable to exercise
* IQ >90
* ADHD

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Reaction time (RT) of mental rotation tasks | 8 weeks
  The experiment involved simultaneously presenting children with two pictures of "giraffes". The image on the left was fixed as the target, and the image on the right showed angle or mirror differences. The angular disparities were 0°, 60°, 120° or 180°. Through rotation, the children were asked to determine, as quickly and accurately as possible, whether the two images were identical.
Reaction time (RT) of modified Stroop task | 8 weeks
  The computerized modified Stroop task includes the following two conditions: a naming (non-execution) and execution condition. In the naming condition, the screen will display a colored "XXX" and the children need to press the key corresponding to the color. In the execution condition, the stimulus will show a distracting-colored word, similar to the classic Stroop, showing Chinese characters in either blue or red; in this test, the children need to press the key corresponding to the color of the word, rather than the meaning of the Chinese character. When the color of the word is consistent with its meaning, the condition is congruent; when the color of the word is inconsistent with its meaning, it is the condition is incongruent.
Standing broad jump | 8 weeks
  The SBJ test, which is completed on a flat surface, is used to evaluate the explosive strength of the lower limbs.
50m sprint | 8 weeks
  The 50m sprint test requires students to start in a standing position and complete a 50m sprint with all their strength. The test is conducted twice, and the fastest result is recorded.
50m*8 shuttle run | 8 weeks
  children are required to run back and forth between two points as quickly as possible.
Safety and Tolerability | 8 weeks
  There were no safety and adverse events

SECONDARY OUTCOMES:
Height | 8 weeks
  Height was measured to the nearest 0.1 cm (Shanghe SH-200G, China)
Weight | 8 weeks
  weight was measured to the nearest 0.1 kg using a portable stadiometer (Shanghe SH-200G, China).

OTHER OUTCOMES:
Safety and Tolerability | From enrollment until at least 12 weeks after completion of study treatment
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai University of Medicine and Health Sciences, Shanghai, Pudong, China

IPD SHARING:
Plan to Share IPD: Undecided
This experiment is still in progress as other research and can be made public at the appropriate time.